CLINICAL TRIAL: NCT03076307
Title: Correlation of Procedural Motor Skills Impairment and 123I-FP-CIT SPECT Uptake in Patients With Early Parkinson's Disease: a Case-control Study
Brief Title: DAT SPECT and Procedural Motor Skills in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Nicolas Nicastro, Dr. Med. Nicolas NICASTRO, University Hospital, Geneva
Allocation: Non-Randomized | Model: Parallel | Purpose: Basic Science
Other Study IDs: CCER 2016-01469
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parkinson's disease (Experimental)
  Interventions: Behavioral: Procedural Motor Skills with mirror-drawing of figures
- Control group (Active Comparator)
  Interventions: Behavioral: Procedural Motor Skills with mirror-drawing of figures

INTERVENTIONS:
Behavioral: Procedural Motor Skills with mirror-drawing of figures — Evaluation of error rate and speed for completion of a procedural motor task

SUMMARY:
Patients with Parkinson's disease (PD) are known to be affected by subtle cognitive impairment early in the disease course, mostly in the executive field. Procedural motor skills, mainly controlled by the basal ganglia associative loop (in particular dorsal caudate nucleus) (Rodriguez-Oroz et al., 2009), have also been studied in patients with PD (Schnider et al., 1995; Muslimovic et al., 2007; Terpening et al., 2013). However, the correlation of dopaminergic 123I-FP-CIT SPECT imaging and cognitive impairment has not been assessed. One reason is the absence of reference values for striatal uptake until recently. Last year, the investigators established local uptake reference values for DAT imaging based on a large cohort of subjects with non-degenerative conditions (Nicastro et al., 2016) and can therefore use these values to precisely assess uptake loss in patients with PD.

With the present study, the investigators expect to enroll patients with early PD for whom a 123I-FP-CIT SPECT has been previously performed in the center. Subjects will perform a specific motor task based on mirror-drawing of star-shaped figures. This will be done by inverting the direction of horizontal/vertical computer mouse movements on the screen. Speed and error rates will be assessed for patients as well as healthy control subjects. Correlation with striatal SPECT uptake, especially caudate nucleus uptake, will be analyzed for PD patients. In addition, resting-state EEG will be performed for all subjects. General medication and dopaminergic drugs in particular, whenever used, will not be discontinued. For all subjects enrolled in the study, cognitive and neurological examination will be performed.

ELIGIBILITY:
Inclusion criteria for PD group:

* Age > 18 year-old
* Diagnosis of PD with onset <2 years from enrollment
* Available DAT SPECT performed in Geneva University Hospitals <6 months before inclusion

Inclusion criteria for control group:

Age- and sex-matched control patients

* Age > 18 year-old
* No known neurological condition interfering with motor and cognitive abilities
* No medication interfering with central nervous system (including antidepressants, antipsychotics, hypnotics)

Exclusion criteria for both groups:

* Major depressive state (Hospital Anxiety and Depression scale ≥11 for depression score)
* Cognitive decline (Mini-Mental Score ≤ 22/30)
* Debilitating tremor (Movement Disorders Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III - rest, postural and action tremor ≥2/4)
* Significant akinesia (MDS-UPDRS III hand brady-akinesia score ≥2/4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Procedural motor performance (error and time) in PD group | 2 days
  Evaluation of error rate and speed for completion of mirror-drawing of star-shaped figures

SECONDARY OUTCOMES:
Resting state EEG connectivity in PD and control groups | 2 days
  Evaluation of resting state EEG connectivity in both groups
Difference >20% in error rate and speed improvement in control and PD groups | 2 days
  Evaluation of a >20%-difference between PD and control groups in terms of speed and error rate for the successive procedural motor task trials

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Neurorehabilitation, Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No